CLINICAL TRIAL: NCT02114177
Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Investigate the Efficacy and Safety of a 12- or 8-Week Treatment Regimen of Simeprevir in Combination With Sofosbuvir in Treatment-Naïve and -Experienced Subjects With Chronic Genotype 1 Hepatitis C Virus Infection Without Cirrhosis
Brief Title: Efficacy and Safety Study of Simeprevir in Combination With Sofosbuvir in Participants With Chronic Hepatitis C Virus Infection Without Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103430; TMC435HPC3017 (Other: Janssen Infectious Diseases BVBA)
Record Dates: First submitted 2014-04-02; First posted 2014-04-15 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C Virus Infection; Simeprevir; Sofosbuvir; HCV; Cirrhosis
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — Simeprevir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Simeprevir/Sofosbuvir) (Experimental): 150 participants will receive 1 capsule of 150 mg simeprevir and 1 tablet of 400 mg sofosbuvir orally (by mouth) once daily for 12 weeks.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir
- Arm 2 (Simeprevir/Sofosbuvir) (Experimental): 150 participants will receive 1 capsule of 150 mg simeprevir and 1 tablet of 400 mg sofosbuvir orally once daily for 8 weeks.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Simeprevir — 150 participants will receive 1 capsule of 150 mg simeprevir orally once daily for 12 weeks in Arm 1.
  Arms: Arm 1 (Simeprevir/Sofosbuvir)
Drug: Simeprevir — 150 participants will receive 1 capsule of 150 mg simeprevir orally once daily for 8 weeks in Arm 2
  Arms: Arm 2 (Simeprevir/Sofosbuvir)
Drug: Sofosbuvir — 150 participants will receive 1 tablet of 400 mg sofosbuvir orally once daily for 12 weeks in Arm 1.
  Arms: Arm 1 (Simeprevir/Sofosbuvir)
Drug: Sofosbuvir — 150 participants will receive 1 tablet of 400 mg sofosbuvir orally once daily for 8 weeks in Arm 2.
  Arms: Arm 2 (Simeprevir/Sofosbuvir)

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of a treatment regimen of 12 weeks or 8 weeks of simeprevir in combination with sofosbuvir in chronic hepatitis C virus (HCV) genotype 1 infected men and women without cirrhosis who are HCV treatment-naïve or treatment-experienced.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), open-label (all people know the identity of the intervention), multicenter study. The study will consist of a screening phase up to 6 weeks, open-label treatment phase of 8 weeks or 12 weeks, and post-treatment follow up phase up to 24 weeks after end of treatment. Approximately 300 participants will be randomly allocated in a 1:1 ratio to receive 150 mg simeprevir in combination with 400 mg sofosbuvir once daily either for 12 weeks (Arm 1) or 8 weeks (Arm 2). Safety evaluations will include assessment of adverse events, clinical laboratory tests, vital signs, and physical examination. The maximum study duration for each participant will be approximately 42 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus (HCV) genotype 1a or 1b infection confirmed before randomization
* Documentation of the presence or absence of a NS3 Q80K polymorphism in HCV genotype 1a infected participants before randomization
* Documentation of the IL28B genotype before randomization
* HCV ribonucleic acid level greater than 10,000 IU/mL at screening
* Treatment-experienced participants must have at least 1 documented previous course of interferon-based regimen with or without ribavirin
* Absence of cirrhosis in participants

Exclusion Criteria:

* Evidence of clinical hepatic decompensation (history or current evidence of ascites, bleeding varices or hepatic encephalopathy)
* Infection/co-infection with HCV non-genotype 1a or 1b
* Co-infection with human immunodeficiency virus (HIV) type 1 or type 2 (HIV-1 or HIV-2) (positive HIV-1 or HIV-2 antibodies test at screening)
* Co-infection with hepatitis-B virus (hepatitis-B-surface-antigen positive)
* Previously been treated with any direct acting anti-HCV agent (approved or investigational) for chronic HCV infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (40):
- United States (38):
  - Dothan, Alabama
  - Bakersfield, California
  - Chula Vista, California
  - Los Angeles, California
  - San Diego, California
  - Englewood, Colorado
  - Bradenton, Florida
  - Jacksonville, Florida
  - Lauderdale Lakes, Florida
  - Maitland, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Marietta, Georgia
  - Indianapolis, Indiana
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Hillsborough, New Jersey
  - Vineland, New Jersey
  - Manhasset, New York
  - New York, New York
  - Asheville, North Carolina
  - Winston-Salem, North Carolina
  - Pittsburgh, Pennsylvania
  - East Greenwich, Rhode Island
  - Providence, Rhode Island
  - Greer, South Carolina
  - Germantown, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Norfolk, Virginia
- Canada (2):
  - Vancouver, British Columbia
  - Montreal, Quebec

REFERENCES:
- [Derived] Kwo P, Gitlin N, Nahass R, Bernstein D, Etzkorn K, Rojter S, Schiff E, Davis M, Ruane P, Younes Z, Kalmeijer R, Sinha R, Peeters M, Lenz O, Fevery B, De La Rosa G, Scott J, Witek J. Simeprevir plus sofosbuvir (12 and 8 weeks) in hepatitis C virus genotype 1-infected patients without cirrhosis: OPTIMIST-1, a phase 3, randomized study. Hepatology. 2016 Aug;64(2):370-80. doi: 10.1002/hep.28467. Epub 2016 Mar 22. PMID 26799692

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 310 participants were randomly allocated to the 2 treatment arms. All participants received at least 1 dose of study drug and were included in intent to treat (ITT) analysis set.
Groups:
- Simeprevir and Sofosbuvir for 8 Weeks: Participants received 1 capsule of 150 milligram (mg) simeprevir and 1 tablet of 400 mg sofosbuvir orally (by mouth) once daily for 8 weeks.
- Simeprevir and Sofosbuvir for 12 Weeks: Participants received 1 capsule of 150 mg simeprevir and 1 tablet of 400 mg sofosbuvir orally (by mouth) once daily for 12 weeks.
Period: Overall Study
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Started | 155 | 155
Completed | 146 | 151
Not Completed | 9 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks | Total
Number analyzed (Participants) | 155 | 155 | 310
Age, Continuous [Median (Full Range); unit: years] | 56 [21 to 70] | 56 [19 to 70] | 56 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 73 | 141
  Male | 87 | 82 | 169

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Sustained Virologic Response 12 Weeks After the Actual End of Treatment (SVR12)
Description: Participants considered to have achieved SVR12, if the hepatitis C virus ribonucleic acid (HCV RNA) is less than (<) lower limit of quantification (LLOQ; 25 international unit per milliliter [IU/mL]) detectable or undetectable at 12 weeks after the actual end of study drug treatment.
Time Frame: 12 weeks after the end of treatment (EOT) (Week 20 or Week 24)
Population: Intent-to-treat (ITT) population included all the randomized participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 155 | 155
Percentage of participants | 82.6 [76.3 to 88.9] | 96.8 [93.7 to 99.9]

2. Secondary Outcome: Percentage of Participants Achieving a Sustained Virologic Response 4 Weeks After the Actual End of Treatment (SVR4)
Description: Participants considered to have achieved SVR4, if the hepatitis C virus ribonucleic acid (HCV RNA) is less than (<) lower limit of quantification (LLOQ; 25 international unit per milliliter [IU/mL]) detectable or undetectable at 4 weeks after the actual end of study drug treatment.
Time Frame: 4 weeks after the end of treatment (EOT) (Week 12 or Week 16)
Population: Intent-to-treat (ITT) population included all the randomized participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 155 | 155
Percentage of Participants | 83.9 [77.8 to 90.0] | 96.8 [93.7 to 99.9]

3. Secondary Outcome: Percentage of Participants Achieving a Sustained Virologic Response 24 Weeks After the Actual End of Treatment (SVR24)
Description: Participants considered to have achieved SVR24, if the hepatitis C virus ribonucleic acid (HCV RNA) is less than (<) lower limit of quantification (LLOQ; 25 international unit per milliliter [IU/mL]) detectable or undetectable at 24 weeks after the Actual end of study drug treatment.
Time Frame: 24 weeks after the end of treatment (EOT) (Week 32 or Week 36)
Population: Intent-to-treat (ITT) population included all the randomized participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 155 | 155
Percentage of participants | 82.6 [76.3 to 88.9] | 96.8 [93.7 to 99.9]

4. Secondary Outcome: Percentage of Participants Achieving a On-treatment Virologic Response
Description: Ontreatment virologic response was determined by HCV RNA results satisfying a specified threshold. <LLOQ undetectable was considered as threshold at any time point. The LLOQ value is 25 IU/mL. EOT=End of Treatment.
Time Frame: Day 14, Day 28, End of treatment (Week 8 or Week 12)
Population: The ITT population included all the randomized participants who took at least 1 dose of study drug. Here, 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 155 | 155
Percentage of participants
  Day 14: < 100 IU/mL (n=154, 152) | 90.9 | 93.4
  Day 14: < 25 IU/mL (n=154, 152) | 77.92 | 79.6
  Day 14: < 25 IU/mL detectable (n=154, 152) | 40.26 | 45.4
  Day 14: < 25 IU/mL undetectable (n=154, 152) | 37.66 | 34.2
  Day 28: < 100 IU/mL (n=154, 153) | 100 | 100
  Day 28: < 25 IU/mL (n=154, 153) | 98.7 | 98.7
  Day 28: < 25 IU/mL detectable (n=154, 153) | 16.2 | 11.1
  Day 28: < 25 IU/mL undetectable (n=154, 153) | 82.5 | 87.6
  EOT: < 100 IU/mL (n=155, 155) | 100 | 100
  EOT: < 25 IU/mL (n=155, 155) | 100 | 100
  EOT: < 25 IU/mL undetectable (n=155, 155) | 100 | 100

5. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Percentage of participants with greater than 1 log10 IU/mL increase in plasma Hepatitis C virus ribonucleic acid level from the lowest level reached (ie, lowest value measured in between baseline and current value), or a confirmed plasma HCV RNA level of greater than 100 IU/mL in participants whose plasma HCV RNA had previously been less than 25 IU/mL.
Time Frame: Up to Week 24
Population: The ITT population included all the randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 155 | 155
Percentage of participants | 0 | 0

6. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Percentage of participants who did not achieve sustained virologic response 12, have less than 25 IU/mL undetectable plasma HCV RNA at end of treatment, and greater than or equal to 25 IU/mL plasma HCV RNA during the follow-up phase.
Time Frame: Up to Week 24
Population: The ITT population included all the randomized participants who took at least 1 dose of study drug. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 155 | 154
Percentage of participants | 17.4 | 2.6

7. Secondary Outcome: Change From Baseline in Hepatitis C Symptom and Impact Questionnaire 4 (HCV-SIQv4) Overall Body System Score (OBSS)
Description: HCVSIQv4 OBSS was a self-administered questionnaire that contained 33 items: 29 questions developed to assess severity or frequency of symptoms associated with HCV or its treatment, 3 questions regarding the impact of symptoms on work/school attendance, and 1 question regarding the impact of symptoms on daily activities. A symptom severity score (the mean of responses to the 29 symptom items); each symptom score was transformed to have a range from 0 to 100 (most severe). Higher HCV SIQv4 scores indicates worse symptom severity, more time missed from work/school, and more impairment in daily activities, respectively.
Time Frame: Baseline (Day 1), Week 4, Week 8, Week 12, Follow-up Week 4, Follow-up Week 12 and Follow-up Week 24
Population: The ITT population included all the randomized participants who took at least 1 dose of study drug. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure and 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 146 | 153
units on a scale
  Baseline (n=145, 149) | 10.8 (0.94) | 13.3 (1.01)
  Change at Week 4 (n=145, 146) | -0.4 (0.83) | -0.9 (0.89)
  Change at Week 8 (n=144, 146) | -0.2 (1.06) | -0.4 (0.90)
  Change at Week 12 (n=0, 141) | NA (NA) — The treatment duration for this Arm is 8 weeks. | 0.1 (0.97)
  Change at Follow-up Week 4 (n=142, 148) | -3.5 (0.88) | -3.0 (0.91)
  Change at Follow-up Week 12 (n=141, 145) | -2.0 (0.86) | -3.5 (0.96)
  Change at Follow-up Week 24 (n=133, 143) | -3.6 (0.99) | -4.4 (0.90)

8. Secondary Outcome: Change From Baseline in Fatigue Severity Scale (FSS) Score up to Follow-up Week 24
Description: The FSS was a self-administered questionnaire with 9 items developed to assess disabling fatigue that has been used extensively in studies of chronic HCV infection. Item responses were measured on a 7point Likert scale ranging from strongly disagree (1 point) to strongly agree (7 points). The 9 items were averaged to produce a total score; a lower total score indicates less severe fatigue. FSS scores have a range from 1 to 7 where higher scores indicate more severe fatigue.
Time Frame: Baseline (Day 1), Week 4, Week 8, Week 12, Follow-up Week 4, Follow-up Week 12 and Follow-up Week 24
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 146 | 153
units on a scale
  Baseline (n=144, 149) | 2.9 (0.13) | 3.2 (0.14)
  Change at Week 4 (n=142, 142) | -0.1 (0.09) | -0.1 (0.13)
  Change at Week 8 (n=142, 144) | -0.1 (0.11) | -0.2 (0.14)
  Change at Week 12 (n=0, 140) | NA (NA) — The treatment duration for this Arm is 8 weeks. | -0.1 (0.15)
  Change at Follow-up Week 4 (n=141, 148) | -0.4 (0.12) | -0.4 (0.13)
  Change at Follow-up Week 12 (n=140, 145) | -0.5 (0.11) | -0.4 (0.15)
  Change at Follow-up Week 24 (n=132, 143) | -0.6 (0.13) | -0.5 (0.14)

9. Secondary Outcome: Change From Baseline in Center for Epidemiologic Studies Depression Scale (CES-D) Scores
Description: The CES-D scale assesses how often during the past week participants experienced 20 symptoms commonly associated with major depression. CES-D scores range from 0 (no symptoms) to 60 (all 20 symptoms most or all of the time during the past 5-7 days). The CES-D scores between 16 and 23 points indicate mild to moderate depressive illness while CES-D scores greater than or equal to 23 indicate probable major depressive illness.
Time Frame: Baseline (Day 1), Week 4, Week 8, Week 12, Follow-up Week 4, Follow-up Week 12 and Follow-up Week 24
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 146 | 153
units on a scale
  Baseline (n=144, 149) | 8.8 (0.72) | 10.2 (0.71)
  Change at Week 4 (n=139, 140) | -0.6 (0.67) | -0.8 (0.52)
  Change at Week 8 (n=141, 144) | -0.6 (0.73) | -0.3 (0.66)
  Change at Week 12 (n=141, 144) | NA (NA) — The treatment duration for this Arm is 8 weeks. | 1.0 (0.72)
  Change at Follow-up Week 4 (n=141, 148) | -2.6 (0.64) | -0.6 (0.68)
  Change at Follow-up Week 12 (n=140, 145) | -1.5 (0.62) | -0.1 (0.72)
  Change at Follow-up Week 24 (n=131, 143) | -2.8 (0.72) | -1.0 (0.70)

10. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension (EQ-5D) Visual Analogue Scale
Description: The EQ-5D questionnaire is a brief, generic health-related quality of life assessment (HRQOL) that can also be used to incorporate participant preferences into health economic evaluations. The EQ-5D questionnaire assesses HRQOL in terms of degree of limitation on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and as overall health using a "thermometer" visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health). Lower scores indicate worsening.
Time Frame: Baseline (Day 1), Week 4, Week 8, Week 12, Follow-up Week 4, Follow-up Week 12 and Follow-up Week 24
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Number analyzed (Participants) | 146 | 153
units on a scale
  Baseline (N=144, 149) | 79.3 (1.53) | 76.7 (1.48)
  Change at Week 4 (n=142, 141) | 4.6 (1.31) | 2.4 (1.05)
  Change at Week 8 (n=142, 144) | 4.0 (1.21) | 2.7 (0.93)
  Change at Week 12 (n=0, 140) | NA (NA) — The treatment duration for this Arm is 8 weeks. | 2.5 (1.14)
  Change at Follow-up Week 4 (n=141, 148) | 6.9 (1.34) | 4.4 (1.12)
  Change at Follow-up Week 12 (n=138, 145) | 5.5 (1.27) | 3.9 (1.37)
  Change at Follow-up Week 24 (n=131, 143) | 6.2 (1.51) | 5.3 (1.28)

ADVERSE EVENTS:
Time Frame: Baseline to End of Treatment (week 8 or week 12)
Description: The total number of adverse events listed in the "Other (nonSerious) Adverse Event" table are based on at least 5 percent of participants experiencing the adverse event in any treatment arm
Arm/Group | Simeprevir and Sofosbuvir for 8 Weeks | Simeprevir and Sofosbuvir for 12 Weeks
Serious Adverse Events (participants affected / at risk) | 3/155 | 2/155
Other Adverse Events (participants affected / at risk) | 68/155 | 65/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simeprevir and Sofosbuvir for 8 Weeks (N=155) | Simeprevir and Sofosbuvir for 12 Weeks (N=155)
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Mania (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simeprevir and Sofosbuvir for 8 Weeks (N=155) | Simeprevir and Sofosbuvir for 12 Weeks (N=155)
Nausea (Gastrointestinal disorders) | 14 | 23
Diarrhoea (Gastrointestinal disorders) | 12 | 11
Constipation (Gastrointestinal disorders) | 8 | 9
Headache (Nervous system disorders) | 26 | 22
Fatigue (General disorders) | 24 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 9
Insomnia (Psychiatric disorders) | 10 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.